CLINICAL TRIAL: NCT01837420
Title: A Randomized, Double Blind, Dose Ranging, Placebo Controlled Study to Evaluate the Efficacy and Safety of Oral VB-201 in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of VB-201 in Patients With Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VB-201-079
Record Dates: First submitted 2012-12-01; First posted 2013-04-23 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — 1-palmityl-2-(4-carboxybutyl)-sn-glycero-3-phosphocholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo with crossover to VB-201 160mg (Other): Subjects on placebo will crossover to VB-201 160 at week 16.
  Interventions: Drug: VB-201 160mg; Drug: Placebo
- VB-201 80mg (Experimental): Subjects will receive VB-201 80mg/day for 24 weeks
  Interventions: Drug: VB-201 80mg
- VB-201 160mg (Experimental): Subjects will received 80mg twice daily for 24 weeks
  Interventions: Drug: VB-201 160mg

INTERVENTIONS:
Drug: VB-201 80mg
  Arms: VB-201 80mg
Drug: VB-201 160mg
  Arms: Placebo with crossover to VB-201 160mg; VB-201 160mg
Drug: Placebo
  Arms: Placebo with crossover to VB-201 160mg

SUMMARY:
This study will examine the safety and efficacy in subjects with moderate to severe psoriasis, as measured by Psoriasis Area and Severity Index(PASI), Body Surface Area (BSA), Dermatology Life Quality Index (DLQI) and other assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, ≥18 to ≤75 years of age, who have a diagnosis of chronic plaque psoriasis for at least 6 months prior to screening;
* Plaque psoriasis covering between 10% to 30 % of body surface area (BSA);
* PASI severity moderate to severe, scoring at least 10 but no higher than 20.

Exclusion Criteria:

* The subject presents with psoriasis that is predominantly guttate, erythrodermic, inverse, pustular or palmo-plantar or an unstable form of psoriasis;
* Previously failed (due to lack of efficacy) treatment with at least one systemic biologic agent for psoriasis (e.g. ustekinumab, adalimumab, etanercept, etc);
* The subject has not undergone wash-out periods of sufficient duration for the following treatments at Baseline: Topical psoriasis treatments: 2 weeks; Systemic (non-biologic) psoriasis treatments: 4 weeks or 5 half-lives (whichever is longer); Biologic psoriasis treatments: 8 weeks or 5 half lives (whichever is longer); Phototherapy: 4 weeks;
* The subject anticipates getting enough ultra-violet light during the study (e.g. sunbathing; tanning salon, etc.) to cause psoriasis to improve;
* History of cancer, with the exception of skin cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
PASI 50 | Week 16 and Week 24
  The proportion of subjects in the VB-201 160 mg (80 mg BID) treatment group who achieve at least 50% improvement from the baseline PASI score at Weeks 16 and 24 (PASI 50) compared to the proportion of PASI 50 responders in the placebo group.

SECONDARY OUTCOMES:
PASI 75 | Week 16 and Week 24
  Proportion of subjects in each of the VB-201 treatment groups and in the combined (both dose groups) VB-201 treatment groups who achieve at least 75% improvement from the baseline PASI score (PASI 75) at Weeks 16 and 24 compared to the proportion of PASI 75 responders in the placebo group.

OTHER OUTCOMES:
Frequency of Adverse Events | From Baseline through safety follow up at Week 28
  As measured by changes from baseline in physical exam, vital signs, ECG, concomitant medications, laboratory values.
Body Surface Area | Week 16 and Week 24
  Change in affected Body Surface Area (BSA) from baseline to Week 16 and Week 24 in each of the VB-201 treatment groups and in the combined (both dose groups) VB-201 treatment groups compared to placebo.
Physician Global Assessment | Week 16 and Week 24
  Change in PGA scores from baseline to Weeks 16 and 24 in each of the VB-201 treatment groups and in the combined (both dose groups) VB-201 treatment groups compared to the placebo group.
Patient Psoriasis Global Assessment | Week 16 and Week 24
  Change in Patient Psoriasis Global Assessment scores from baseline to Weeks 16 and 24 in each of the VB-201 treatment groups and in the combined (both dose groups) VB-201 treatment groups compared to the placebo group.
PASI 50- 80 mg/ day | Week 16 and Week 24
  The proportion of subjects in the VB-201 80 mg/day treatment group who achieve at least 50% improvement from the baseline PASI score at Weeks 16 and 24 (PASI 50) compared to the proportion of PASI 50 responders in the placebo group.
Change in PASI score | Week 16 and Week 24
  The mean change in the PASI score from baseline to Weeks 16 and 24 in each of the two VB-201 treatment groups and in the combined (both dose groups) VB-201 treatment groups compared to the mean change in the placebo group.
Itching Visual Analogue Scale | Week 16 and Week 24
  Change in itching VAS from baseline to weeks 16 and 24 in each of the VB 201 treatment groups and in the combined (both dose groups) VB-201 treatment groups compared to placebo.
Pain Visual Analogue Scale | Week 16 and Week 24
  Change in pain VAS from baseline to weeks 16 and 24 in each of the VB 201 treatment groups and in the combined (both dose groups) VB-201 treatment groups compared to placebo.
Dermatology Life Quality Index | Week 16 and Week 24
  Change in the DLQI scores from baseline to Weeks 16 and 24 in each of the VB 201 treatment groups and in the combined (both dose groups) VB-201 treatment groups compared to placebo.

CONTACTS AND LOCATIONS:
Locations (4):
- VBL Investigative Site, Kiel, Germany
- VBL Investigative Site, Netanya, Israel
- VBL Investigative Site, Warsaw, Poland
- VBL Investigative Site, Barcelona, Spain